CLINICAL TRIAL: NCT05226390
Title: Safety, Reactogenicity and Immunogenicity of a Novel MVA-SARS-2-ST Vaccine Candidate Administered as Inhalation Boost in SARS-CoV-2 Immunized Adults - Phase I Study
Brief Title: Safety, Reactogenicity and Immunogenicity of a Novel MVA-SARS-2-ST Vaccine Candidate
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: cohort could not be recruited
Sponsor: Hannover Medical School (Other)
Collaborators: German Center for Infection Research (Other); IDT Biologika (Unknown); Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MVA-S2-S-R01
Record Dates: First submitted 2022-01-31; First posted 2022-02-07 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: COVID-19 Vaccines
Keywords: MVA-SARS-COV-2; MVA-SARS-2-ST

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 x 107 IU/dose MVA-SARS-2-ST (Experimental): All Participants will receive a single booster dose of 1 x 107 IU MVA-SARS-2-ST in 0.5 mL as inhalation (total inhaled volume 0.5 mL)
  Interventions: Biological: MVA-SARS-2-ST

INTERVENTIONS:
Biological: MVA-SARS-2-ST — In this trial MVA-SARS-2-ST will be used. Each vial contains 1 x 107 IU/dose MVA-SARS-2-ST in 0.5 mL as active ingredient. The solution will be used for nebulization and direct administration to the respiratory tract.

SUMMARY:
This will be a phase I, single-center trial, including a total of 30 participants in two cohorts.

Cohort 1 (n=6): Healthy male or female adults aged 18 - ≤ 60 previously primary immunized with two vaccinations with any regimen using any EU marketed SARS-CoV-2 vaccine (mRNA-, vector-, protein-based, attenuated SARS-CoV-2 virus) or with a single application of COVID-19 Vaccine Janssen.

Cohort 2 (n=24): Healthy male or female adults aged 18 - ≤ 60 primary immunized with two vaccinations with any regimen using any EU marketed SARS-CoV-2 vaccine (mRNA-, vector-, protein-based, attenuated SARS-CoV-2 virus) or with a single application of COVID-19 Vaccine Janssen and subsequently booster immunized with any EU marketed mRNA vaccine

Both cohorts will be assigned to inhaled vaccination with MVA-SARS-2-ST

ELIGIBILITY:
Inclusion Criteria:

The subject must not be enrolled before all inclusion criteria (including test results) are confirmed. Subjects meeting all of the criteria listed below will be included in the study.

1. Signed written informed consent from subject prior to any study-related procedure and willingness to comply with treatment and follow-up procedures
2. Healthy men or women, aged ≥ 18 ≤ 60 at day of inclusion having received either

   1. primary immunization (cohort 1) with any regimen using any EU marketed SARS- CoV-2 vaccine or
   2. subsequently booster immunization (cohort 2) with any EU marketed mRNA vaccine

   at least 3 months prior to enrollment
3. Adults with SARS-CoV-2 specific IgG concentration between 10 RU/ml and 1200 RU/ml determined by Anti-SARS-CoV-2-QuantiVac-ELISA (IgG)
4. Males or non-pregnant, non-lactating females of child-bearing potential with negative pregnancy test at screening who agree to comply with the applicable contraceptive requirements of the protocol (Section 3.4) from at least 14 days prior to vaccination and during the entire duration of the study.

   or

   Females without child-bearing potential defined as follows:
   * at least 6 weeks after surgical sterilization by bilateral tubal ligation or bilateral oophorectomy or
   * hysterectomy or uterine agenesis or
   * ≥ 50 years and in postmenopausal state > 1 year or
   * < 50 years and in postmenopausal state > 1 year with serum FSH > 40 IU/l and serum estrogen < 30 ng/l or a negative estrogen test, both at screening
5. Normal pulmonary function: FEV1 predicted ≥ 80% and FEV1/FVC > 70%
6. Body mass index 18.5 - 30.0 kg/m2 and weight > 50 kg at screening
7. Subject is capable of understanding the investigational nature, potential risks and benefits of the clinical trial

Exclusion Criteria:

Subjects are excluded from the study if any of the following criteria are met at screening or on dosing day.

1. Previous MVA or rMVA vaccination
2. Known allergy to the components of the SARS-CoV-2 vaccine product as chicken proteins or history of life-threatening reactions to vaccine containing the same substances
3. Known history of anaphylaxis to vaccination or any allergy likely to be exacerbated by any component of the trial vaccine
4. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance; safety laboratory screening evaluation can be repeated a maximum of two times
5. Any finding in the medical history and physical examination deviating from normal and assessed as clinically relevant by the investigator
6. Evidence in the subject's medical history or in the medical examination that might influence the absorption, distribution, metabolism or excretion of the investigational medicinal product
7. Current smoking/ vaping or smoking /vaping in the previous year.
8. Clinically relevant findings in ECG
9. Any confirmed or suspected immunosuppressive or immunodeficient condition, cytotoxic therapy in the previous 5 years, and/or diabetes
10. Asthma, chronic obstructive pulmonary disease or other lung disease
11. Respiratory tract infection in the 4 weeks prior to study treatment
12. Any chronic or active neurologic disorder, including seizures, and epilepsy, excluding a single febrile seizure as a child
13. Known intolerance to medication used during bronchoscopy, i.e. midazolam and lidocaine.
14. Treatment with ß-adrenoceptor antagonists
15. Alcohol abuse (consumption of more than 20 g per day for females and 30 g per day for males)
16. Drug abuse or positive drug screening
17. Any positive result for HIV1/2, HCV antibody or HBs antigen testing
18. Moderate or severe illness and/or fever >38 °C within 1 week prior to vaccination
19. History of blood donation within 60 days of enrollment or plans to donate within the treatment phase
20. Participation in a clinical trial or use of an investigational product within 30 days or five times the half-life of the investigational product -whichever is longer- prior to receiving the first dose within this study
21. Investigator or employee of the study site or Sponsor with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, natural or adopted child) of the investigator or employee with direct involvement in the proposed study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
The nature, frequency and severity of adverse events associated with MVA-SARS-2-ST | day 0
  Occurrence of solicited local reactogenicity signs and symptoms
The nature, frequency and severity of adverse events associated with MVA-SARS-2-ST | day 1
  Occurrence of solicited local reactogenicity signs and symptoms
The nature, frequency and severity of adverse events associated with MVA-SARS-2-ST | day 2
  Occurrence of solicited local reactogenicity signs and symptoms
The nature, frequency and severity of adverse events associated with MVA-SARS-2-ST | day 3
  Occurrence of solicited local reactogenicity signs and symptoms
The nature, frequency and severity of adverse events associated with MVA-SARS-2-ST | day 4
  Occurrence of solicited local reactogenicity signs and symptoms
The nature, frequency and severity of adverse events associated with MVA-SARS-2-ST | day 5
  Occurrence of solicited local reactogenicity signs and symptoms
The nature, frequency and severity of adverse events associated with MVA-SARS-2-ST | day 6
  Occurrence of solicited local reactogenicity signs and symptoms
The nature, frequency and severity of adverse events associated with MVA-SARS-2-ST | day 7
  Occurrence of solicited local reactogenicity signs and symptoms
Change from baseline of pulmonary function associated with MVA-SARS-2-ST | day 0 (2h), day 1, 3, 7, 14, 28, 56, 140
  Change from baseline of pulmonary function measured by spirometry as forced vital capacity (FVC) (%)
Change from baseline of pulmonary function associated with MVA-SARS-2-ST | day 0 (2h), day 1, 3, 7, 14, 28, 56, 140
  Change from baseline of pulmonary function measured by spirometry as forced expiratory volume in 1 second (FEV1) (%)
Change from baseline of pulmonary function associated with MVA-SARS-2-ST | day 0 (2h), day 1, 3, 7, 14, 28, 56, 140
  Change from baseline of pulmonary function measured by spirometry as FEV1/FVC (%)
Change from baseline of pulmonary function associated with MVA-SARS-2-ST | day 0 and twice daily on days 1, 2, 3, 4, 5, 6, 7
  Change from baseline of pulmonary function measured by peak flow as peak expiratory flow (PEF) frequently
Occurrence of solicited systemic reactogenicity signs and symptoms associated with MVA-SARS-2-ST | day 0
  Occurrence of solicited systemic reactogenicity signs and symptoms vaccination
Occurrence of solicited systemic reactogenicity signs and symptoms associated with MVA-SARS-2-ST | day 1
  Occurrence of solicited systemic reactogenicity signs and symptoms vaccination
Occurrence of solicited systemic reactogenicity signs and symptoms associated with MVA-SARS-2-ST | day 2
  Occurrence of solicited systemic reactogenicity signs and symptoms vaccination
Occurrence of solicited systemic reactogenicity signs and symptoms associated with MVA-SARS-2-ST | day 3
  Occurrence of solicited systemic reactogenicity signs and symptoms vaccination
Occurrence of solicited systemic reactogenicity signs and symptoms associated with MVA-SARS-2-ST | day 4
  Occurrence of solicited systemic reactogenicity signs and symptoms vaccination
Occurrence of solicited systemic reactogenicity signs and symptoms associated with MVA-SARS-2-ST | day 5
  Occurrence of solicited systemic reactogenicity signs and symptoms vaccination
Occurrence of solicited systemic reactogenicity signs and symptoms associated with MVA-SARS-2-ST | day 6
  Occurrence of solicited systemic reactogenicity signs and symptoms vaccination
Occurrence of solicited systemic reactogenicity signs and symptoms associated with MVA-SARS-2-ST | day 7
  Occurrence of solicited systemic reactogenicity signs and symptoms vaccination
Occurrence of unsolicited adverse events (AE) associated with MVA-SARS-2-ST | from day 0 to day 28 after vaccination
  Occurrence of unsolicited adverse events (AE)
Change of safety laboratory measures associated with MVA-SARS-2-S | day 1, 3, 7, 14, 28, 56, 140
  Change from baseline of safety laboratory measures
Occurrence of serious adverse events (SAE) associated with MVA-SARS-2-ST | through study completion, an average of 5 month
  Occurrence of serious adverse events (SAE)

SECONDARY OUTCOMES:
To evaluate immunogenicity of the candidate MVA-SARS-2-ST | day 7, 14, 28, 56 and 140
  Change from baseline of levels of binding antibodies against SARS-CoV-2 spike S1 protein measured by ELISA in blood
To evaluate immunogenicity of the candidate MVA-SARS-2-ST | day 14
  Change from baseline of levels of binding antibodies against SARS-CoV-2 spike S1 protein measured by ELISA in (bronchial alveolar lavage) BAL on day 14

CONTACTS AND LOCATIONS:
Overall Officials: Jens Hohlfeld, Prof., Principal Investigator — Hannover Medical School, Department of Respiratory Medicine and Fraunhofer ITEM, Division of Clinical Airway Research; Reinhold Förster, Prof., Study Chair — Hannover Medical School Institute of Immunology
Locations (1):
- Hannover Medical School ZKS - Early Clinical Trial Unit at CRC Hannover, Hanover, Germany

IPD SHARING:
Plan to Share IPD: No